CLINICAL TRIAL: NCT00865137
Title: An Open-label, Single-centre Study to Assess the Effect of Food on the Relative Bioavailability of Orally Administered Tacrolimus Modified Release Formulation, FK506E (MR4), in Stable Kidney Transplant Recipients
Brief Title: An Open Study Assessing Bioavailability of a Modified Formulation of Tacrolimus in Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FG-506E-04-32; EudraCT No.: 2005-005714-20
Record Dates: First submitted 2009-03-16; First posted 2009-03-19 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Pharmacokinetics; Tacrolimus modified release; FK506E
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 FK506E (Experimental)
  Interventions: Drug: Tacrolimus, modified release

INTERVENTIONS:
Drug: Tacrolimus, modified release — Oral
  Other Names: FK506E; MR4; Advagraf; Prograf XL

SUMMARY:
The purpose of this study is to evaluate the effect of food on the oral bioavailability of tacrolimus modified release (MR4) capsules together with a standard continental breakfast. The objective is to assess the pharmacokinetics and relative bioavailability with and without food.

DETAILED DESCRIPTION:
Stable kidney transplant recipients who are participating in the clinical trial FG-506-14-02 and who are currently being treated with FK506E (MR4) under fasted conditions and who have had no changes in any of their medications for at least seven days will be enrolled in the sub-study. Following enrolment, all patients will remain on all their medication and the same dosing regimen throughout the study.During the study two 24 hour blood concentration time profiles will be collected, each one on the last day of Period 2 and Period 3 of the sub-study as follows:

Profile 1 on Day 7 under fasted conditions

Profile 2 on Day 14 under non-fasted conditions

A total of five scheduled visits are planned.

At least 24 patients with two complete, evaluable profiles are needed to estimate the effect of food on the oral bioavailability of FK506E (MR4).

Blood sampling - For each sample a 2 mL aliquot of whole blood will be collected. The total blood volume for the two profiles taken per patient will be approximately 40 mL.

ELIGIBILITY:
Inclusion Criteria:

* Stable kidney transplant patient aged ≥ 18 years who is participating in clinical trial FG-506-14-02 and is being treated with FK506E (MR4)
* The total daily dose of each immunosuppressive medication, including FK506E (MR4), or any other concomitant medication has remained unchanged for at least seven days prior to enrolment
* Patient has a serum creatinine level < 265 μmol/L at enrolment
* Female patient of childbearing potential must have a negative serum or urine pregnancy test prior to enrolment and must have agreed to practice effective birth control during the study

Exclusion Criteria:

* Patient had previously received an organ transplant other than kidney
* Patient with any form of substance abuse, psychiatric disorder or condition which may complicate communication with the investigator
* Patient had experienced any rejection episode within 90 days prior to enrolment, any rejection episode within the last six months that had required anti-lymphocyte antibody therapy or more than two rejection episodes within the last 12 months
* Patient has a chronic dysfunction of the kidney
* Patient had major changes in her/his immunosuppressive regimen within the last three months prior to enrolment
* Patient has significant liver disease, defined as having elevated SGPT/ALT and/or SGOT/AST and/or total bilirubin levels (at least two times the upper value of the normal range at the investigational site) during the 28 days prior to enrolment
* Patient receives insulin therapy
* Patient requires treatment with medication or substances known to interfere with tacrolimus metabolism or having taken such medication within 28 days prior to enrolment and during participation
* Patient had any unstable medical condition that could interfere with the study
* Patient is pregnant or a breast-feeding mother
* Patient is known to be positive for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Assess pharmacokinetic parameters | Day 7 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Maastricht, Netherlands